CLINICAL TRIAL: NCT04752553
Title: Pros and Cons of Telemedicine in Diagnosis and Management
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Heba A Yassa (Other)
Responsible Party: Sponsor-Investigator, Heba A Yassa, Professor of Forensic Medicine and Clinical Toxicology, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AssiutU1234
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: the Study Focus on the Uses of Telephone and Other New Technology in Medicine, Diagnosis and Treatment
Keywords: Telemedicine - malpractice - telehealth
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Telemedicine "healing at a distance" Telemedicine has many advantages especially in time of pandemics for both doctors and patients, low cost and easily accessibility. Pandemics especially COVID 19 has radically change the medical team thoughts about the telemedicine. It can decrease the exposure of the medical team to infection and expected by some of the medical team to be very beneficial if done in good and legal manner. Although, telemedicine has many advantages, also has many disadvantages and medicolegal problems, breakdown in the relationship between medical teams and patients, mis diagnosis or wrong treatment. There are many legal and ethical aspects of telemedicine.

DETAILED DESCRIPTION:
Telemedicine "healing at a distance" Telemedicine has many advantages especially in time of pandemics for both doctors and patients, low cost and easily accessibility. Pandemics especially COVID 19 has radically change the medical team thoughts about the telemedicine. It can decrease the exposure of the medical team to infection and expected by some of the medical team to be very beneficial if done in good and legal manner. Although, telemedicine has many advantages, also has many disadvantages and medicolegal problems, breakdown in the relationship between medical teams and patients, mis diagnosis or wrong treatment. There are many legal and ethical aspects of telemedicine. These include the medical responsibilities, the confidentiality and privacy of the patients can not be maintained, the jurisdictional problems. Shortage of medical practitioners and specialists, shortage of internet facilities, low education levels in some patients all are problems facing the telemedicine in developing countries. The evolution of telemedicine poses a series of legal problems ranging from the profiles on the subject of authorization and accreditation to those concerning the protection of patient confidentiality, the definition and solution of which, in the absence of specific regulatory provisions, is mainly left to the assessment of compatibility of the practices adopted so far, with the general regulatory framework.

This research will be done to clarify the role of telemedicine, and if it has a share hand or the upper hand if compared with traditional medicine.

ELIGIBILITY:
Inclusion Criteria:

* doctors of all specialty
* Patients
* police man and who work in law

Exclusion Criteria:

* No exclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all population can be included in the study
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-08-10 (Estimated); Study Completion 2022-02-10 (Estimated)

PRIMARY OUTCOMES:
- To provide an overview about the pros and cons of the telemedicine in Egypt especially in the period of the COVID 19 pandemic. | 6 months
  describe the pros and cons of the telemedicine
- To assess the impact of telehealth on clinical outcomes from the view of the doctors, patients. | 6 months
  list the impact of telehealth and telemedicine on doctors and patients

SECONDARY OUTCOMES:
- To evaluate the opinion of the law and the malpractice problems that can face doctors due to the use of telemedicine. | one year
  List the law opinion about the telemedicine

CONTACTS AND LOCATIONS:
Locations (1):
- heba Yassa, Asyut, Egypt

REFERENCES:
- [Background] Ferorelli D, Nardelli L, Spagnolo L, Corradi S, Silvestre M, Misceo F, Marrone M, Zotti F, Mandarelli G, Solarino B, Dell'Erba A. Medical Legal Aspects of Telemedicine in Italy: Application Fields, Professional Liability and Focus on Care Services During the COVID-19 Health Emergency. J Prim Care Community Health. 2020 Jan-Dec;11:2150132720985055. doi: 10.1177/2150132720985055. PMID 33372570
- [Background] Durupt M, Bouchy O, Christophe S, Kivits J, Boivin JM. [Telemedicine in rural areas: general practitioners' representations and experiences]. Sante Publique. 2016 Oct 19;28(4):487-497. French. PMID 28155753
- [Background] Ateriya N, Saraf A, Meshram VP, Setia P. Telemedicine and virtual consultation: The Indian perspective. Natl Med J India. 2018 Jul-Aug;31(4):215-218. doi: 10.4103/0970-258X.258220. PMID 31134926
- [Background] Vidal-Alaball J, Acosta-Roja R, Pastor Hernandez N, Sanchez Luque U, Morrison D, Narejos Perez S, Perez-Llano J, Salvador Verges A, Lopez Segui F. Telemedicine in the face of the COVID-19 pandemic. Aten Primaria. 2020 Jun-Jul;52(6):418-422. doi: 10.1016/j.aprim.2020.04.003. Epub 2020 Apr 17. PMID 32402477
- See also: http://pubmed.ncbi.nlm.nih.gov/32643663/ — http://pubmed.ncbi.nlm.nih.gov/32643663/